CLINICAL TRIAL: NCT06002776
Title: Our Anesthesia Experiences in Hepatopancreatobiliary Surgery Practices: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Gokce, Assistant Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Sisli Hamidiye Etfal TRH
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Experience, Life
Keywords: major abdominal surgery; Revised Cardiac Risk Index; Epidural analgesia; perioperative fluid management; ERAS protocols

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative and perioperative anaesthetic management: We have planned to retrospectively review data for patients aged 18 and above who underwent major abdominal surgery at our center between October 2017 and February 2022. The study aims to record data regarding the administration of thromboprophylaxis, preoperative hemoglobin values, and Revised Cardiac Risk Index scores and their impact on one-year postoperative mortality. Additionally, we intend to examine the effects of the amount of fluid administered during the perioperative period, the application of epidural analgesia, and the use of blood products on hospital stay duration and one-year postoperative mortality.
  Interventions: Other: a retrospective study

INTERVENTIONS:
Other: a retrospective study — a retrospective study

SUMMARY:
Has the evolving anesthetic management in major abdominal surgeries had a positive impact on patients' one-year postoperative mortality and length of hospital stay? Which of the anesthetic management parameters have influenced mortality and hospital stay duration in these patients? To address these questions, we have planned to retrospectively review patients who underwent surgery at our center.

DETAILED DESCRIPTION:
In our study, we aimed to compile our practices over the last 5 years by evaluating the impact of perioperative and postoperative anesthetic management on morbidity and mortality in hepatopancreatobiliary surgical patients. Our primary outcome was to form a comprehensive understanding of our anesthesia experiences during the preoperative, perioperative, and postoperative periods in this patient group. Our secondary outcome was to assess the influence of preoperative and perioperative anesthetic management on the morbidity and mortality of these patients.

ELIGIBILITY:
Inclusion Criteria:

* The study will include data from patients who have undergone their first operation with the diagnoses of liver malignancy, cholangiocarcinoma, and pancreatic malignancy during the period from October 2017 to February 2022.

Exclusion Criteria:

* Data from patients who were deemed inoperable during the perioperative period after being taken into surgery with their current diagnosis, as well as data from patients who underwent repeat operations, were excluded from the study for their second and subsequent hospitalizations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: data from all patients aged 18 and above who underwent major abdominal surgery with diagnoses of liver malignancy, cholangiocarcinoma, and pancreatic malignancy
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
form a comprehensive understanding of our anesthesia experiences during the preoperative, perioperative, and postoperative periods in this patient group | october2017-february2022

SECONDARY OUTCOMES:
assess the influence of preoperative and perioperative anesthetic management on the morbidity and mortality of these patients. | october2017-february2022

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training and Researching Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All patient data will be kept confidential.

REFERENCES:
- [Background] Snowden C, Prentis J. Anesthesia for hepatobiliary surgery. Anesthesiol Clin. 2015 Mar;33(1):125-41. doi: 10.1016/j.anclin.2014.11.008. Epub 2014 Dec 31. PMID 25701932
- [Background] Hemmerling TM. Pain management in abdominal surgery. Langenbecks Arch Surg. 2018 Nov;403(7):791-803. doi: 10.1007/s00423-018-1705-y. Epub 2018 Oct 3. PMID 30284029
- [Background] von der Forst M, Weiterer S, Dietrich M, Loos M, Lichtenstern C, Weigand MA, Siegler BH. [Perioperative fluid management in major abdominal surgery]. Anaesthesist. 2021 Feb;70(2):127-143. doi: 10.1007/s00101-020-00867-7. German. PMID 33034685